CLINICAL TRIAL: NCT04650126
Title: A Phase I, Randomized, Double-blind, Parallel Group and Placebo-controlled Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Atrosimab in Response to Single Ascending Intravenous Infusion Doses.
Brief Title: Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Atrosimab (ATM001) in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Baliopharm Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATM001-001
Record Dates: First submitted 2020-11-05; First posted 2020-12-02 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2021-07

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATM001 (Experimental): Escalating dose levels of ATM001 administered as single dose in healthy subjects
  Interventions: Biological: ATM001
- ATM001 Placebo (Placebo Comparator): Escalating dose levels of ATM001 Placebo administered as single dose in healthy subjects
  Interventions: Biological: ATM001 Placebo

INTERVENTIONS:
Biological: ATM001 — monovalent anti-TNF-receptor 1 antibody format
  Other Names: Atrosimab
  Arms: ATM001
Biological: ATM001 Placebo — ATM001 Placebo
  Arms: ATM001 Placebo

SUMMARY:
This is a double-blind, parallel group and placebo-controlled clinical study to assess safety tolerability, pharmacokinetics and pharmacodynamics of Atrosimab in healthy volunteers

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* body mass index 18-32 kg/m2
* normal physical examination, clinical laboratory values and ECG
* additional inclusion criteria apply

Exclusion Criteria:

* febrile or infectious illness at least 7 days prior to the first administration
* any active physical disease, acute or chronic
* history of alcohol or drug abuse
* history of chronic or recurrent metabolic, renal, hepatic, pulmonary, gastrointestinal, neurological, endocrinological, immunological, psychiatric, or cardio-vascular disease, myopathies and bleeding tendency
* additional exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-07-12 (Actual); Primary Completion 2022-03-24 (Actual); Study Completion 2022-03-24 (Actual)

PRIMARY OUTCOMES:
pharmacokinetic (PK): Area under the analyte concentration-time curve from time 0 and extrapolated to infinite time (AUC 0-∞) | 8 days
PK: Area under the plasma concentration curve from administration until the last quantifiable sampling point (AUC 0-t) | 8 days
PK: Maximum Plasma Concentration [Cmax] | 8 days
PK: Terminal half life (t1/2) | 8 days
PK: Apparent terminal elimination rate constant (λz) | 8 days
PK: Mean residence time (MRT) | 8 days
PK: Clearance (CL) | 8 days
PK: Apparent volume of distribution (Vz) | 8 days
Any adverse event, serious adverse event (SAE) | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kristi McLendon, MD, Principal Investigator — Q-Pharm Pty Limited
Locations (1):
- Q-Pharm, Herston, Brisbane, Australia